CLINICAL TRIAL: NCT01624948
Title: Safety and Efficacy of Mycophenolic Acid Withdrawal With Conversion to Zortress (Everolimus) in Renal Transplant Recipients With BK Virus Infection
Brief Title: Safety and Efficacy Study of Everolimus to Treat BK Virus Infection in Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001AUS184T
Record Dates: First submitted 2012-06-15; First posted 2012-06-21 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-07

CONDITIONS: BK Virus Infection
Keywords: BK virus; Kidney Transplantation; Immunologic Monitoring
MeSH Terms: interventions — Everolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Everolimus+Tacrolimus/Prednisone (Experimental): This arm (group 1) will undergo mycophenolic acid (MPA) discontinuation with the addition of Zortress (everolimus) to their current regimen of tacrolimus and prednisone; All patients in group 1 will receive Zortress (everolimus) at a starting dose of 0.75 mg PO b.i.d. (1.5 mg/day). Everolimus whole blood trough levels will be monitored at pre-specified time points to achieve a range of 3-8 ng/mL. Group 1 patients will continue on prednisone and tacrolimus with a target whole blood trough level of 3-6 ng/mL.
  Interventions: Drug: Everolimus
- Standard of care: 50% reduction of MPA (Active Comparator): This arm (group 2) patients will continue with tacrolimus (target trough level of 6-10 ng/mL), prednisone, and undergo a 50% reduction of the MPA dose, which is the standard immunosuppression treatment for renal transplant recipients with evidence of BKV infection. At months 1, 2, and 3 post-randomization urine and plasma BKV levels will be re-checked. Renal allograft biopsies will be done for cause as clinically indicated.
  Interventions: Drug: Mycophenolic acid dose reduction

INTERVENTIONS:
Drug: Everolimus — Everolimus will be administered orally at a starting dose of 0.75 mg PO b.i.d. (1.5 mg/day). Everolimus whole blood trough levels will be monitored at pre-specified time points to achieve a range of 3-8 ng/mL. Group 1 patients will continue on prednisone and tacrolimus with a target whole blood trough level of 3-6 ng/mL.
  Other Names: Zortress
  Arms: Everolimus+Tacrolimus/Prednisone
Drug: Mycophenolic acid dose reduction — Group 2 patients will undergo a 50% reduction of the mycophenolic acid (MPA) dose, and continue with tacrolimus (target trough level of 6-10 ng/mL), and prednisone.
  Other Names: CellCept; Myfortic
  Arms: Standard of care: 50% reduction of MPA

SUMMARY:
This study is examining the safety and efficacy of converting anti-rejection therapy from mycophenolic acid (MPA) to Zortress (everolimus) in renal transplant recipients with BK virus infection.

The study will also determine if immune monitoring tests can detect an association between BK virus infection and transplant rejection episodes, based on the specific BKV infection treatment regimen.

The investigators hypothesize that an anti-rejection regimen with Zortress (everolimus) and tacrolimus + prednisone will be superior to a standard regimen of reduced dose MPA and tacrolimus + prednisone in patients who have undergone renal transplantation and have active BKV infections.

DETAILED DESCRIPTION:
This is a pilot study designed as a single center, randomized, open-label trial study comparing the safety and efficacy of MPA discontinuation with the addition of Zortress (everolimus) versus standard immunosuppression reduction in adult patients who have undergone a renal transplant and who have evidence of BKV infection. All kidney transplant recipients at University of California, San Francisco (UCSF) are screened for BKV in the urine and plasma at months 1, 3, 6, 9, and 12 post-transplantation. The presence of viruria > 1 million copies/mL and/or viremia prompts a 50% reduction in the MPA dose as well as monthly monitoring of BKV in the urine and plasma. Renal transplant patients found to have BK viruria > 1 million copies/mL and/or viremia > 500 copies/mL on any screening lab will be eligible for enrollment.

Before any study-related evaluations are performed, the patient must give written informed consent. Once consent is obtained, patients will be randomized in consecutive blocks of 10, such that there will be 5 patients allocated to each group for each block. Only the study coordinator will have access to the block sequences. Patients will be randomized to one of two groups: group 1 will undergo MPA discontinuation with the addition of Zortress (everolimus) to their current regimen of tacrolimus and prednisone; group 2 will undergo a 50% dose reduction in MPA and continue with tacrolimus and prednisone.

The two groups will be as follows: All patients in group 1 will undergo discontinuation of MPA and will receive Zortress (everolimus) at a starting dose of 0.75 mg PO b.i.d. (1.5 mg/day). Everolimus whole blood trough levels will be monitored at pre-specified time points to achieve a range of 3-8 ng/mL. Group 1 patients will continue on prednisone and tacrolimus with a target whole blood trough level of 3-6 ng/mL. Group 2 patients will continue with tacrolimus (target trough level of 6-10 ng/mL), prednisone, and undergo a 50% reduction of the MPA dose. At months 1, 2, and 3 post-randomization urine and plasma BKV levels will be re-checked. Renal allograft biopsies will be done for cause as clinically indicated. Tacrolimus trough levels are lower in the Zortress (everolimus) arm in order to minimize any potential nephrotoxicity with this drug combination as well as minimize the risk of over-immunosuppression.

In all patients, routine transplant monitoring labs will be performed monthly as part of standard of care including a measurement of blood urea nitrogen (BUN) and creatinine (Cr), complete blood count (CBC), tacrolimus trough levels, urine protein excretion and fasting lipids.

During the 3 month treatment period patients will be seen in clinic at baseline and months 1, 2, and 3 for follow-up. The assessment to address the primary objective will be performed at the end of the treatment period (Month 3). An interim analysis will be performed once 50% enrollment is reached.

In a sub-group of patients (30 patients total; 15 in group 1 and 15 in group 2) using our whole-blood assay measuring p70S6 kinase phosphorylation, the investigators will investigate the correlation between inhibition of p70S6 kinase phosphorylation with BKV replication. Finally, by measuring both p70S6 phosphorylation inhibition as well as expression of the nuclear factor of activated T cells (NFAT)-regulated genes Interleukin (IL)-2, interferon gamma and GM-CSF, the investigators will correlate rejection episodes in patients maintained on lower immunosuppression alone versus those on a Zortress (everolimus) -based regimen. As patients are assigned to their intervention group based on the randomization scheme they will be offered enrollment in this sub-group analysis. All patients will be sequentially enrolled in the sub-group analysis until the 30 subject goal is reached with 15 subjects per group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female renal transplant recipients 18-75 years of age (primary or re-transplant)
* Recipients of cadaveric, living unrelated or living related donor kidney
* Baseline immunosuppression (IS) consisting of tacrolimus, MPA, and prednisone
* Patients with BK viruria ≥ 1 million copies/mL and/or viremia (> 500 copies/mL) found on routine BKV screening.
* Patients who have given written informed consent to participate in the study

Exclusion Criteria:

* Patients who are ABO incompatible transplants
* Patients with an abnormal liver profile such as Alanine Aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, or total bilirubin > 3x ULN at the time of randomization
* Patients with severe total hypercholesterolemia (> 350 mg/dL) or total hypertriglyceridemia (> 500 mg/dL). Patients on lipid lowering drugs with controlled hyperlipidemia are acceptable.
* Patients with a platelet count < 100,000/mm3 at randomization
* Patients with an ANC < 1,500/mm3 or WBC < 4.5mm3
* Patients with a known hypersensitivity to the study drug or to drugs of similar chemical classes.
* Patients being treated with drugs (other than tacrolimus) that are potent inducers or inhibitors of cytochrome P4503A4
* Patients who have any surgical or medical condition, such as severe diarrhea, active peptic ulcer disease, or uncontrolled DM, which, in the opinion of the investigators, might significantly alter the absorption, distribution, metabolism and/or excretion of study medication.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive urine human chorionic gonadotrophin laboratory test
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, UNLESS they are using two birth control methods. The two methods can be a double barrier method or a barrier method plus a hormonal method.
* Adequate barrier methods of contraception include: diaphragm, condom (by the partner), intrauterine device (copper or hormonal), sponge or spermicide. Hormonal contraceptives include any marketed contraceptive agent that includes an estrogen and/or a progestational agent.
* Reliable contraception should be maintained throughout the study and for 7 days after study drug discontinuation.
* Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL and estradiol < 20 pg/mL] or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
* Patients with baseline urine protein excretion > 500mg/day
* Patients with Estimated Glomerular Filtration Rate (eGFR) < 40 ml/min
* Patients who have undergone desensitization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2015-02 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Webber, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Wajih Z, Karpe KM, Walters GD. Interventions for BK virus infection in kidney transplant recipients. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD013344. doi: 10.1002/14651858.CD013344.pub2. PMID 39382091

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: 50% Reduction of Mycophenolic Acid (MPA): This arm (group 2) patients will continue with tacrolimus (target trough level of 6-10 ng/mL), prednisone, and undergo a 50% reduction of the MPA dose, which is the standard immunosuppression treatment for renal transplant recipients with evidence of BK polyomavirus (BKV) infection. At months 1, 2, and 3 post-randomization urine and plasma BKV levels will be re-checked. Renal allograft biopsies will be done for cause as clinically indicated.
  Mycophenolic acid dose reduction: Group 2 patients will undergo a 50% reduction of the mycophenolic acid (MPA) dose, and continue with tacrolimus (target trough level of 6-10 ng/mL), and prednisone.
Period: Overall Study
Arm/Group | Everolimus+Tacrolimus/Prednisone | Standard of Care: 50% Reduction of Mycophenolic Acid (MPA)
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Everolimus+Tacrolimus/Prednisone: This arm (group 1) will undergo MPA discontinuation with the addition of Zortress (everolimus) to their current regimen of tacrolimus and prednisone; All patients in group 1 will receive Zortress (everolimus) at a starting dose of 0.75 mg PO b.i.d. (1.5 mg/day). Everolimus whole blood trough levels will be monitored at pre-specified time points to achieve a range of 3-8 ng/mL. Group 1 patients will continue on prednisone and tacrolimus with a target whole blood trough level of 3-6 ng/mL.
  Everolimus: Everolimus will be administered orally at a starting dose of 0.75 mg PO b.i.d. (1.5 mg/day). Everolimus whole blood trough levels will be monitored at pre-specified time points to achieve a range of 3-8 ng/mL. Group 1 patients will continue on prednisone and tacrolimus with a target whole blood trough level of 3-6 ng/mL.
- Standard of Care: 50% Reduction of Mycophenolic Acid (MPA): This arm (group 2) patients will continue with tacrolimus (target trough level of 6-10 ng/mL), prednisone, and undergo a 50% reduction of the MPA dose, which is the standard immunosuppression treatment for renal transplant recipients with evidence of BKV infection. At months 1, 2, and 3 post-randomization urine and plasma BKV levels will be re-checked. Renal allograft biopsies will be done for cause as clinically indicated.
  Mycophenolic acid dose reduction: Group 2 patients will undergo a 50% reduction of the mycophenolic acid (MPA) dose, and continue with tacrolimus (target trough level of 6-10 ng/mL), and prednisone.
- Total: Total of all reporting groups
Arm/Group | Everolimus+Tacrolimus/Prednisone | Standard of Care: 50% Reduction of Mycophenolic Acid (MPA) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (10.3) | 49.9 (12.4) | 52.18 (11.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 13 | 11 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 11 | 15 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Donor Type [Number; unit: participants]
  Living | 7 | 8 | 15
  Standard Deceased | 11 | 10 | 21
  ECD | 2 | 2 | 4
Transplant Number [Number; unit: participants]
  First | 16 | 17 | 33
  Second | 4 | 3 | 7
Etiology of End Stage Renal Disease (ESRD) [Number; unit: participants]
  Diabetes | 2 | 4 | 6
  Hypertension | 3 | 3 | 6
  GN | 12 | 11 | 23
  Other | 3 | 2 | 5
Calculated Panel Reactive Antibodies (cPRA) [Mean (Standard Deviation); unit: Percentage of Potential Donors] — The Calculated Panel Reactive Antibodies (cPRA) represents the percentage of potential donors that will be preemptively declined due to the presence of one or more unacceptable antigens. CPRA is a computer calculation based upon HLA frequencies derived from the US donor population and the risk they attribute to circulating antibodies in a candidate's serum directed against those specific HLA antigens.
  Percentage of Potential Donors | 14.4 (28.8) | 25.5 (36.3) | 19.93 (32.82)
Ureteral Stent at Transplant [Number; unit: participants]
  Ureteral Stent Present | 0 | 2 | 2
  No Ureteral Stent Present | 20 | 18 | 38
Renal Graft Function [Number; unit: participants] — Delayed Graft Function was defined as > or =1 dialysis session during the first week posttransplant
  participants
    Delayed Graft Function | 6 | 2 | 8
    Normal Graft Function | 14 | 18 | 32

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Reduction of BK Viruria and/or Clearance of BK Viremia
Description: composite outcome of a 50% or greater reduction in BKV urine levels and/or complete clearance of BKV viremia by 3 months after randomization
Time Frame: 3 months post-randomization
Measure: Number; unit: participants
Arm/Group | Everolimus+Tacrolimus/Prednisone | Standard of Care: 50% Reduction of MPA
Number analyzed (Participants) | 20 | 20
participants | 11 | 8
Statistical Analysis 1: Comparison: Everolimus+Tacrolimus/Prednisone vs Standard of Care: 50% Reduction of MPA; Test type: Superiority or Other; p = 0.53, Fisher Exact

2. Secondary Outcome: Evaluation for the Development of BK Virus Nephropathy or Doubling of BK Viremia Levels
Description: A doubling of BK viremia levels or the development of BKV nephropathy in subjects enrolled in the experimental study arm will prompt a conversion to standard care therapy. We will closely monitor BKV levels in the urine and blood and assess renal function monthly, as per our usual standard of care. Based on BKV results as well as renal function, as assessed by serum Cr, biopsies may be done for cause. Patients will have a final visit at month 4 to monitor for adverse events.
Time Frame: 3 months post-randomization
Measure: Number; unit: participants
Arm/Group | Everolimus+Tacrolimus/Prednisone | Standard of Care: 50% Reduction of MPA
Number analyzed (Participants) | 20 | 20
participants | 2 | 2

3. Secondary Outcome: p70S6 Kinase Phosphorylation
Time Frame: 3 months post-randomization
Population: 19 patients enrolled in the immune-monitoring subset; 1 participant did not have a 3-month assay.
Measure: Median (95% Confidence Interval); unit: Mean Fluorescence Intensity
Groups:
- Reached Primary Endpoint: >50% reduction of BKV viruria and/or clearance of BKV viremia
Arm/Group | Reached Primary Endpoint | Failed to Reach Primary Endpoint
Number analyzed (Participants) | 6 | 12
Mean Fluorescence Intensity | 5002 [1821 to 8389] | 4353 [2676 to 6442]
Statistical Analysis 1: Comparison: Reached Primary Endpoint vs Failed to Reach Primary Endpoint; Difference in p70S6 kinase phosphorylation as measured by mean fluorescence intensity (MFI) between those patients who reached the primary endpoint and those who did not; Test type: Superiority or Other; p = 0.67, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Cholesterol
Time Frame: 3 months post-randomization
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Everolimus+Tacrolimus/Prednisone | Standard of Care: 50% Reduction of MPA
Number analyzed (Participants) | 20 | 20
mg/dL | 212 (56.8) | 170 (29.8)
Statistical Analysis 1: Comparison: Everolimus+Tacrolimus/Prednisone vs Standard of Care: 50% Reduction of MPA; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Proteinuria
Time Frame: 3 months post-randomization
Measure: Mean (Standard Deviation); unit: g/g creatinine
Arm/Group | Everolimus+Tacrolimus/Prednisone | Standard of Care: 50% Reduction of MPA
Number analyzed (Participants) | 20 | 20
g/g creatinine | 0.16 (.1) | 0.23 (.21)

6. Secondary Outcome: Median Between the Calculated Mean Residual Expression of NFAT-regulated Genes
Description: Measurement of the expression of three NFAT-regulated genes IL-2, interferon gamma, and GM-CSF, to predict a rejection episode.
  The residual gene expression after Tacrolimus intake was calculated as T1.5/T0*100, where T0 is the adjusted number of transcripts at Tacrolimus pre-dose level and T1.5 is the number of transcripts 1.5 hours after drug intake. For all three genes the residual expression was averaged and presented as "MRE of NFAT-regulated genes."
Time Frame: 3 months post-randomization
Population: a subset of 19 participants enrolled in the immune-monitoring portion of the study
Measure: Median (95% Confidence Interval); unit: percent residual expression
Groups:
- Rejection: Any biopsy-proven rejection episode
- No Rejection: No biopsy-proven rejection episode
Arm/Group | Rejection | No Rejection
Number analyzed (Participants) | 3 | 16
percent residual expression | 46.35 [-16 to 94.82] | 29.12 [20.83 to 41.34]
Statistical Analysis 1: Comparison: Rejection vs No Rejection; Test type: Superiority or Other; p = 0.49, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Groups:
- Everolimus+Tacrolimus/Prednisone: Everolimus: MPA discontinuation with the addition of Zortress (everolimus) to current regimen of tacrolimus and prednisone; Zortress (everolimus) at a starting dose of 0.75 mg PO b.i.d. (1.5 mg/day). Everolimus whole blood trough levels monitored at pre-specified time points to achieve a range of 3-8 ng/mL. Continue on prednisone and tacrolimus with a target whole blood trough level of 3-6 ng/mL.
- Standard of Care: 50% Reduction of MPA: Mycophenolic acid dose reduction: continue with tacrolimus (target trough level of 6-10 ng/mL), prednisone, and undergo a 50% reduction of the MPA dose, which is the standard immunosuppression treatment for renal transplant recipients with evidence of BKV infection. At months 1, 2, and 3 post-randomization urine and plasma BKV levels re-checked. Renal allograft biopsies will be done for cause as clinically indicated.
Arm/Group | Everolimus+Tacrolimus/Prednisone | Standard of Care: 50% Reduction of MPA
Serious Adverse Events (participants affected / at risk) | 2/20 | 3/20
Other Adverse Events (participants affected / at risk) | 13/20 | 9/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus+Tacrolimus/Prednisone (N=20) | Standard of Care: 50% Reduction of MPA (N=20)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
CMV Pnemonia/Viremia (Infections and infestations) | 0 (0) | 1 (1)
Acute Cellular Rejection (Grade 1) (Immune system disorders) | 0 (0) | 1 (1)
Anemia and shortness of breath (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sepsis/UTI (Infections and infestations) | 0 (0) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus+Tacrolimus/Prednisone (N=20) | Standard of Care: 50% Reduction of MPA (N=20)
GI Upset (Gastrointestinal disorders) | 2 (2) | 0 (0)
UTI (Infections and infestations) | 2 (2) | 2 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
BK Viremia allograft nephropathy (Infections and infestations) | 2 (2) | 1 (1)
Edema (General disorders) | 1 (1) | 0 (0)
Herpes Simplex 1 Oral Ulcer (Infections and infestations) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Transaminitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acute kidney injury with chest pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Borderline Rejection (Immune system disorders) | 1 (1) | 0 (0)
Insomnia (General disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nightsweats (General disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyperlipidemia (Endocrine disorders) | 2 (2) | 0 (0)
CMV Viremia (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No